CLINICAL TRIAL: NCT02800200
Title: The Long-term Effect of Combined Platelet Rich Plasma With Extracorporeal Shock Wave Therapy in Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Combined PRP and ESWT for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending physician of physical medicine and rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB No: 2-105-05-026
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: platelet rich plasma; extracorporeal shock wave
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Platelet rich plasma (Experimental): The ultrasoud-guided injection with Platelet rich plasma (3cc) was perfomed in both groups.
  Interventions: Procedure: Platelet rich plasma; Device: shock wave
- Active shock wave (Experimental): One-session active shock wave 2 weeks later after PRP injection was performed in intervention group.
  Interventions: Procedure: Platelet rich plasma; Device: shock wave
- Sham shock wave (Placebo Comparator): One-session sham shock wave 2 weeks later after PRP injection was performed in control group.
  Interventions: Procedure: Platelet rich plasma; Device: shock wave

INTERVENTIONS:
Procedure: Platelet rich plasma — Sono-guided injection with 3 cc Platelet rich plasma were performed in both groups.
Device: shock wave — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs).

SUMMARY:
The platelet rich plasma (PRP) and extracorporeal shock wave therapy (ESWT) are new and potential treatment for patients with kinds of musculoskeletal disorders. Although few clinical studies have showed beneficial effect of PRP and ESWT for regeneration of peripheral neuropathy, the effect of combined PRP and ESWT is absent so far.

DETAILED DESCRIPTION:
We perform a prospective randomized, double-blinded study to investigate the combined effect of PRP and ESWT in patients with carpal tunnel syndrome.

Patients were randomized into intervention and control group. Participants in intervention group received sono-guided injection with 3cc PRP and one-session active ESWT and control group received sono-guided injection with 3cc PRP and one-session sham ESWT. The evaluation was performed pretreatment as well as on the 4th, 8th, 12th, 16th and 24 week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 year-old.
2. Typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test, numbness/tingling in at least two of the first, second, or third digits, and in whom the diagnosis was confirmed using an electrophysiological study.

Exclusion Criteria:

1. Cancer
2. Coagulopathy
3. Pregnancy
4. Inflammation status
5. Patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previously undergone wrist surgery or steroid injection for CTS.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area in median nerve on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline of electrophysiological study on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  electrophysiological study according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, School of Medicine, National Defense Medical Center
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Malahias MA, Johnson EO, Babis GC, Nikolaou VS. Single injection of platelet-rich plasma as a novel treatment of carpal tunnel syndrome. Neural Regen Res. 2015 Nov;10(11):1856-9. doi: 10.4103/1673-5374.165322. PMID 26807124
- [Result] Wu YT, Ke MJ, Chou YC, Chang CY, Lin CY, Li TY, Shih FM, Chen LC. Effect of radial shock wave therapy for carpal tunnel syndrome: A prospective randomized, double-blind, placebo-controlled trial. J Orthop Res. 2016 Jun;34(6):977-84. doi: 10.1002/jor.23113. Epub 2015 Dec 10. PMID 26610183